CLINICAL TRIAL: NCT00671190
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Study to Evaluate the Phase-Shifting Effects of Repeated Daily Dosing of Ramelteon in Healthy Subjects
Brief Title: Safety and Efficacy of Ramelteon in Healthy Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-02-TL-375-018; U1111-1114-8304 (Registry Identifier: WHO)
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Sleep Disorder
Keywords: Sleep Disorder; Circadian Rhythm Sleep Disorder; Drug Therapy
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Disorders, Circadian Rhythm | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Ramelteon 1 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Ramelteon 2 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Ramelteon 4 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Ramelteon 8 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 1 mg, tablets, orally once daily for up to 5 days
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 1 mg QD
Drug: Ramelteon — Ramelteon 2 mg, tablets, orally once daily for up to 5 days
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 2 mg QD
Drug: Ramelteon — Ramelteon 4 mg, tablets, orally once daily for up to 5 days
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 4 mg QD
Drug: Ramelteon — Ramelteon 8 mg, tablets, orally once daily for up to 5 days
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 8 mg QD
Drug: Placebo — Ramelteon placebo-matching tablets, orally once daily for up to 5 days
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to determine the phase-advance in circadian rhythms in healthy adults subjects taking ramelteon, once daily (QD).

DETAILED DESCRIPTION:
Circadian rhythms are the innate daily fluctuation of physiologic or behavior functions, included sleep-wake states, generally tied to the 24-hour daily dark-light cycle. Circadian Rhythm Sleep Disorders share a common chronophysiologic basis in which the major feature is a misalignment between the patient's sleep pattern and the sleep pattern that is desired or regarded as the societal norm.

Circadian Rhythm Sleep Disorders affect a sizable portion of the United States population, representing a significant underserved need. It has been estimated that 7% of all adolescents suffer from Delayed Sleep Phase Syndrome. Approximately 1% of all middle-aged people have Advanced Sleep Phase Syndrome. There are 21 million people who are shift workers and between 5% to 20% of these workers develop severe symptoms of Shift Work Sleep Disorder soon after starting shift work. Time Zone Change (Jet Lag) Syndrome can affect millions of travelers each year. Most symptoms are a result of sleep deprivation.

Current treatment of these disorders include behavioral therapy, light therapy and use of hypnotics and stimulants. Melatonin has also been used with mixed results.

The effects of melatonin on circadian phase depend on the time at which it is administered, and are generally opposite those of light. Specifically, melatonin given in the evening results in an advance of the circadian system to an earlier hour ("phase advance"). While melatonin appears to be useful in the treatment of sleep disruption in the blind, the phase shifting ability of native melatonin is much less than that of light, limiting its utility in the treatment of circadian dysfunction in sighted individuals.

Ramelteon is under global development as a sleep-promoting agent. Ramelteon demonstrates affinity and selectivity for human melatonin-1 or melatonin-2 receptors. Ramelteon also demonstrates full agonist activity relative to melatonin in cells expressing human melatonin-1 or melatonin-2 receptors.

The purpose of this study is to determine whether ramelteon given over multiple days can produce a phase advance in circadian rhythms as measured in salivary melatonin levels in dim-light conditions. Participation in this study is anticipated to be about 4 weeks.

ELIGIBILITY:
Inclusion Criteria

* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration
* Habitual bedtime is between 10:00 p.m. and 1:00 a.m.
* Body mass index between 18 and 30, inclusive.
* Medial subjective sleep latency of less than 30 minutes and a median subjective total sleep time of greater than 6.5 but less than 9 hours.

Exclusion Criteria

* Known hypersensitivity to ramelteon or related compounds, including melatonin, and melatonin related compounds.
* Previously participated in a study involving ramelteon.
* Participated in any other investigational study and/or taken any investigational drug within 30 days or five half-lives prior to the first dose of single-blind study medication, whichever is longer.
* Sleep schedule changes required by employment (eg, shift worker) within three months prior to the administration of single-blind study medication.
* Flown across greater than three time zones within 21 days prior to or during screening.
* Participated in a weight loss program or has substantially altered their exercise routine within 30 days prior to the administration of single-blind study medication.
* Ever had a history of seizures, sleep apnea, restless leg syndrome, periodic limb movement syndrome, chronic obstructive pulmonary disease, schizophrenia, bipolar disorder, mental retardation, or cognitive disorder.
* History of primary sleep disorders as determined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised within the past 6 months.
* History of psychiatric disorder (including anxiety or depression) within the past 12 months.
* History of alcohol abuse within the past 12 months, as defined in Diagnostic and Statistical Manual of Mental Disorders, 4th Edition Revised, or regularly consumes more than 14 alcoholic drinks per week, or consumes any alcoholic drinks 2 hours prior to bedtime.
* History of drug abuse within the past 12 months.
* Current neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematologic, or metabolic disease.
* Apnea hypopnea index (per hour of sleep) greater than 10.
* Periodic leg movement syndrome with arousal index (per hour of sleep) greater than 10 as seen on the polysomnography screening night.
* Positive urine drug screen.
* Smokes greater than 3 cigarettes per day or uses tobacco products during nightly awakenings.
* Reports high caffeine consumption (greater than 500 mg daily).
* Any clinically important abnormal finding as determined by a medical history, physical examination, electrocardiogram, or clinical laboratory tests, as determined by the investigator.
* Positive hepatitis panel including anti-hepatitis.
* Unwilling to remain in the sleep laboratory in dim-light conditions for 5 days and nights or fully cooperate with site personnel.
* Any additional condition(s) that in the Investigator's opinion would:

  * affect sleep/wake function
  * prohibit the subject from completing the study
  * not be in the best interest of the subject.
* Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication, including:

  * Anxiolytics
  * Central nervous system active drugs (including herbal)
  * Antipsychotics
  * Narcotic analgesics
  * Antidepressants
  * Beta blockers
  * Anticonvulsants
  * St. John's Wort
  * Sedating H1 antihistamines
  * Kava-kava
  * Systemic steroids
  * Ginkgo-biloba
  * Respiratory stimulants
  * Over the counter and prescription stimulants
  * Decongestants
  * Over-the-counter and prescription diet aids

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2005-03; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Dim Light Melatonin Secretion Offset Time. | Days 1, 2, 3, and 4 or Final Visit.

SECONDARY OUTCOMES:
Dim-Light Melatonin Onset (DLMOn) time. | Days 1, 2, 3, and 4 or Final Visit.

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science, Study Director — Takeda
Locations (13):
- United States (13):
  - Hot Springs, Arkansas
  - Los Angeles, California
  - San Diego, California
  - Miami, Florida
  - Atlanta, Georgia
  - Macon, Georgia
  - Danville, Indiana
  - Overland Park, Kansas
  - Metairie, Louisiana
  - Chevy Chase, Maryland
  - Las Vegas, Nevada
  - Dublin, Ohio
  - Columbia, South Carolina

REFERENCES:
- [Result] Richardson GS, Zee PC, Wang-Weigand S, Rodriguez L, Peng X. Circadian phase-shifting effects of repeated ramelteon administration in healthy adults. J Clin Sleep Med. 2008 Oct 15;4(5):456-61. PMID 18853704
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI